CLINICAL TRIAL: NCT05530343
Title: A Multicenter Randomized Trial of Seattle Biopsy Protocol Versus Wide-Area Transepithelial Sampling in Patients With Barrett's Esophagus Undergoing Surveillance (The SWAT-BE Study)
Brief Title: Seattle Biopsy Protocol Versus Wide-Area Transepithelial Sampling in Patients With Barrett's Esophagus Undergoing Surveillance
Acronym: SWAT-BE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Screening
Other Study IDs: 18-2431
Record Dates: First submitted 2022-09-02; First posted 2022-09-07 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-06

CONDITIONS: Barrett Esophagus; Barretts Esophagus With Dysplasia; Esophageal Adenocarcinoma
Keywords: Barrett's Esophagus; Esophageal Adenocarcinoma; Dysplasia
MeSH Terms: conditions — Barrett Esophagus; Adenocarcinoma Of Esophagus

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Seattle protocol, then WATS3D brushings. (Other): Participants in the screening or surveillance population that receive the Seattle protocol, then WATS3D brushings, during the same procedure.
  Interventions: Diagnostic Test: Seattle protocol; Diagnostic Test: WATS3D brushings
- WATS3D brushings, then Seattle Protocol. (Other): Participants in the screening or surveillance population that receive the WATS3D brushings, then the Seattle protocol, during the same procedure.
  Interventions: Diagnostic Test: Seattle protocol; Diagnostic Test: WATS3D brushings

INTERVENTIONS:
Diagnostic Test: Seattle protocol — Participants undergo 4-quadrant biopsies with standard biopsy forceps taken at 2 cm intervals. For participants undergoing a confirmatory endoscopy for cases in which discordant results are noted (WATS3D positive for dysplasia/cancer and Seattle biopsy negative for dysplasia/cancer), repeat biopsies will be taken at 1 cm intervals along with target biopsies from any visible lesions.
Diagnostic Test: WATS3D brushings — Participants undergo 2 WATS3D biopsies of every 5 cm segment of Barrett's esophagus, starting from the gastroesophageal junction and moving proximally through the entire segment of Barrett's.

SUMMARY:
The purpose of this research study is to learn about the best approach to sample patients with known or suspected Barrett's esophagus (BE) by comparing the standard Seattle biopsy protocol to sampling using wide area transepithelial sampling (WATS3D).

Barrett's esophagus is a common condition that is used to spot patients at increased risk of developing a type of cancer in the esophagus (swallowing tube) called esophageal adenocarcinoma. The 5-year survival rate is as low as 18% for patients who get esophageal adenocarcinoma, but the rate may be improved if the cancer is caught in its early stages. Barrett's esophagus can lead to dysplasia, or precancerous changes, which occurs when cells look abnormal but have not developed into cancer. If the abnormal cells increase from being slightly abnormal (low-grade dysplasia), to being very abnormal (high-grade dysplasia), the risk of developing cancer (esophageal adenocarcinoma) goes up. Therefore, catching dysplasia early is very important to prevent cancer.

Endoscopic surveillance is a type of procedure where endoscopists run a tube with a light and a camera on the end of it down a patients throat and remove a small piece of tissue. The piece of tissue, called a biopsy, is about the size of the tip of a ball-point pen and is checked for abnormal cells and cancer cells.

Patients are being asked to be in this research study because they have been diagnosed with BE or suspected to have BE, and will need an esophagogastroduodenoscopy (EGD).

Patients with BE undergo sampling using the Seattle biopsy protocol during which samples are obtained from the BE in a four quadrant fashion every 2 cm along with target biopsies from any abnormal areas within the BE. Another sampling approach is WATS3D which utilizes brushings from the BE.

While both of these procedures are widely accepted approaches to sampling patients with BE during endoscopy, there is not enough research to show if one is better than the other.

Participants in this study will undergo sampling of the BE using both approaches (Seattle biopsy protocol and WATS-3D); the order of the techniques will be randomized.

Up to 2700 participants will take part in this research. This is a multicenter study involving several academic, community and private hospitals around the country.

DETAILED DESCRIPTION:
Methodology:

Patients with non-dysplastic Barrett's esophagus (BE) undergoing surveillance and patients meeting criteria for screening for BE with columnar-lined esophagus detected at endoscopy will be recruited in this multicenter randomized controlled trial.

All patients will undergo upper endoscopy using high-definition white light endoscopy and electronic chromoendoscopy (NBI/FICE). The findings (detection of visible lesions/abnormal mucosal or vascular pattern) with electronic chromoendoscopy will be recorded.

Patients will be randomized to receive sampling using either the Seattle biopsy protocol or WATS3D. The Seattle protocol will entail obtaining random biopsies every 2 cm in a 4-quadrant fashion. Biopsies will be taken from any visible lesion (no matter how subtle) and will be submitted in separate jars and excluded from the comparative analysis of the study. The WATS3D procedure will be conducted using a standardized protocol. Patients will then receive sampling using the technique to which they were not assigned to by randomization. This allows for all patients to receive standard of care (sampling using the Seattle biopsy protocol), and to determine concordance between the two sampling techniques acknowledging that one sampling technique could potentially affect the results of other sampling technique.

In patients with discordant results (WATS3D positive and random biopsy negative), repeat upper endoscopy with sampling using the Seattle biopsy protocol will be performed in an attempt to confirm the findings noted at WATS3D. This will be performed in the surveillance and screening population. Biopsy specimens will be submitted for histopathologic examination for routine clinical care. For the purpose of this study, all biopsy specimens will be sent to the Cleveland Clinic for interpretation by a central GI pathologist who will be blinded to patient details and to reading by the WATS3D pathologist.

Study Duration:

Interventions performed as described above will be performed during one endoscopic procedure. The endpoints in this study will include progression to dysplasia, cancer, need for endoscopic eradication therapy, and death.

Planned enrollment period: 2.5 years. Planned duration of the study: 3 years.

Study Centers:

To maximize the generalizability of results, this randomized controlled trial will be conducted across different practice settings that include tertiary care centers, closed healthcare networks and large community practices at approximately 14 sites.

Anticipated Number of Participants:

2298 (see Statistical Methodology below)

* 1982 to compare diagnostic yield of dysplasia between the two approaches in BE patients undergoing surveillance
* 316 to compare diagnostic yield of intestinal metaplasia between the two approaches in patients undergoing screening for BE

Statistical Methodology:

For a prospective randomized trial in detecting LGD, HGD or EAC comparing the Seattle protocol, the current standard practice, to wide-area transepithelial sampling (WATS3D) where all positive results for dysplasia or EAC with WATS3D sampling not detected on Seattle biopsy protocol at index endoscopy will require confirmation by repeat sampling using the Seattle biopsy protocol at repeat endoscopy, the following sample sizes were calculated assuming α=0.05 and power of 0.8. All calculations are completed using PROC POWER in SAS 9.4 for Fisher's exact test unless otherwise noted.

For the primary aim (surveillance population), the investigators will compare the proportion of positive results between the Seattle protocol and WATS3D where all positive results for dysplasia or EAC with WATS3D sampling not detected on Seattle biopsy protocol at index endoscopy will require confirmation by repeat sampling using the Seattle biopsy protocol at repeat endoscopy with either Pearson's chi-square test or Fisher's exact test for proportions. Positive findings of dysplasia or EAC on WATS not detected on Seattle biopsy protocol at index endoscopy or subsequent repeat endoscopy with sampling using the Seattle biopsy protocol will not be considered as dysplasia or EAC detected by WATS for the primary analysis. Previous pooled estimates indicated a 2.5% detection rate with Seattle protocol and 4.9% with WATS3D, resulting in a need for 828 participants for each arm (a total of 1656). However, the investigators are restricting to WATS3D cases which are confirmed with target biopsy or Seattle protocol at the initial visit or a follow-up sample when results are discordant. Assuming a 95% confirmation rate, 991 participants are need for each arm to compare a 2.5% detection rate for Seattle protocol and 4.655% for WATS3D (a total of 1982).

For the primary aim (screening population), the investigators will compare the proportion of positive results between techniques to which patients are randomized with Fisher's exact test for proportions. Previous pooled estimates indicated a 40% intestinal metaplasia detection rate with Seattle protocol and 60% with WATS3D. However, the investigators are restricting to WATS3D cases which are confirmed with target biopsy or Seattle protocol at the initial visit or a follow-up sample when results are discordant. Assuming a 95% confirmation rate, 158 participants are need for each arm to compare a 40% detection rate for Seattle protocol and 57% for WATS3D (a total of 316).

The investigators will conduct one interim analysis using Lan and DeMet's alpha spending function approximating O'Brien-Fleming boundaries. Based the sample size estimates above, the investigators expect the interim analysis will occur after the data for 991 participants (50% enrollment) has been collected. This interim analysis will be restricted to the primary aim in the surveillance population. No interim analysis will be conducted to address the primary aim in the screening population. In the case where study enrollment does not stop early due to efficacy, all participating physicians will be blinded to the results of this interim analysis.

As a secondary analysis, the investigators will use results from both the randomized procedure and the follow-up procedure with the protocol to which patients were not randomized to perform a paired analysis of the concordance between the two diagnostic tests. Although an important analysis for determining whether WATS3D could be used instead of the Seattle protocol, due to the risk of the initial biopsy affecting these results of the follow up procedure this is a secondary analysis. Given the sample size of 1982 for the primary outcome, there is greater than 99.9% power to detect a difference in the paired results between proposed discordant proportions of 0.3575% for Seattle protocol positive and WATS3D negative to 3.11% for WATS3D positive and Seattle protocol negative using McNemar's test for paired nominal data. These discordant proportion estimates are derived from prior pooled data for dysplasia detection rates of 4.9% for WATS3D alone and 2.5% for Seattle protocol alone, with the discordant proportions of test results derived from data reported in Vennalaganti assuming that only 80% of WATS3D positive and Seattle protocol negative cases are verified with targeted follow-up biopsies to confirm the diagnosis.

The comparison of yield of dysplasia will also be conducted based on expert pathology review for biopsy and WATS3D specimens. The overall proportion of cases with visible lesions with their associated pathology results will be recorded and will not be a part of the analyses comparing the diagnostic yield of dysplasia between the Seattle biopsy protocol with WATS3D.

The primary outcome comparing diagnostic yield of any dysplasia and intestinal metaplasia between the two randomized arms will use either Pearson's chi-square or Fisher's exact test for portions. The secondary analysis for paired data will use McNemar's test and will exclude cases that were WATS3D positive but could not be confirmed by a concurrent (Seattle protocol) or follow-up endoscopic biopsies using the Seattle biopsy protocol. A sensitivity analysis will be completed which includes WATS3D positive cases that did not have diagnostic confirmation with biopsy. Comparison for the detection of intestinal metaplasia between the two strategies will use McNemar's test for paired data including all cases.

ELIGIBILITY:
Inclusion Criteria:

Surveillance Population

* Undergoing surveillance endoscopy for a diagnosis of non-dysplastic Barrett's esophagus (NDBE, based on last endoscopic procedure; patients with prior history of low-grade dysplasia/indefinite for dysplasia with NDBE at last endoscopy can be included)
* Barrett's esophagus (BE) length of at least M1
* English and Spanish speaking
* Able to comprehend and complete the consent form
* Age18-89 years
* Life-expectancy of at least 2 years

Screening Population

* Undergoing endoscopy for screening of BE
* BE length of at least M1
* English and Spanish speaking
* Able to comprehend and complete the consent form
* Age 18-89 years
* Expected life-expectancy of at least 2 years

Physicians

-All participating sites will include physicians who are trained in the use of WATS3D and certified by the site PI. All endoscopists will need to complete a minimum of three cases to be eligible to participate in the study.

Exclusion Criteria:

Surveillance Population

* BE patients undergoing surveillance or evaluation for endoscopic eradication therapy (EET) for prior diagnosis of BE related dysplasia or esophageal adenocarcinoma (EAC)
* Active erosive esophagitis with LA Grade B or higher
* Esophageal varices
* Prior history of EET
* Prior history of esophageal or gastric surgery, except for uncomplicated fundoplication
* Pregnancy

Screening Population

* BE patients undergoing surveillance or evaluation for EET for prior diagnosis for BE-related dysplasia or EAC
* Active erosive esophagitis with LA Grade B or higher
* Esophageal varices
* Prior history of esophageal or gastric surgery, except for uncomplicated fundoplication
* Pregnancy

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2298 (Estimated)
Dates: Start 2022-10-03 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Diagnostic yield of dysplasia (Surveillance population only) | up to 1 year
  Proportion of positive results between the Seattle protocol and WATS3D technique. Positive results include low-grade dysplasia (LGD), high-grade dysplasia (HGD), and esophageal adenocarcinoma (EAC). All positive results for dysplasia or EAC with WATS3D sampling not detected on Seattle biopsy protocol at index endoscopy will require confirmation by repeat sampling using the Seattle biopsy protocol.
Diagnostic yield of intestinal metaplasia (Screening population only) | up to 1 year
  Proportion of positive results between the Seattle protocol and WATS3D technique. Positive results include intestinal metaplasia. All positive results for intestinal metaplasia/dysplasia or esophageal adenocarcinoma (EAC) with WATS3D sampling not detected on Seattle biopsy protocol at index endoscopy will require confirmation by repeat sampling using the Seattle biopsy protocol.

SECONDARY OUTCOMES:
Detection of intestinal metaplasia (Surveillance population only) | baseline
  Proportion of positive results between the Seattle protocol and WATS3D technique. Positive results include intestinal metaplasia.
Diagnostic yield between the Seattle protocol and WATS3D Vs. the Seattle protocol alone (Surveillance population only) | up to 1 year
  Proportion of positive results of low-grade dysplasia (LGD), high-grade dysplasia (HGD), and esophageal adenocarcinoma (EAC) between the Seattle protocol and WATS3D technique Vs. the WATS3D technique alone. All positive results for intestinal metaplasia/dysplasia or EAC with WATS3D sampling not detected on Seattle biopsy protocol at index endoscopy will require confirmation by repeat sampling using the Seattle biopsy protocol.
Time of procedure as measured by total sampling time (Surveillance population only) | baseline
  Total sampling time for the Seattle protocol is measured by the time the first forceps biopsy was placed into the channel to the time the final forceps biopsy was removed from the channel. Total sampling time for the WATS3D technique is measured by the time the first WATS3D brush was placed into the channel to the time the final WATS3D brush was removed from the channel.
Quality adjusted life years (Surveillance population only) | up to 5 years
  The investigators will conduct a cost-effectiveness analysis between the two sampling techniques using data collected from the randomized control trial (cost for procedures and follow-up, detection of dysplasia or cancer, need for endoscopic eradication therapies, biopsy and pathology costs, complications, among others). The primary endpoint for the cost-effectiveness analysis will be the incremental cost-effectiveness ratio with a predefined willingness to pay off $100k per quality adjusted life years.
Number of patients referred for endoscopic eradication therapy (EET) between Seattle protocol and WATS3D (Surveillance population only) | up to 1 year
  Proportion of patients referred for endoscopic eradication therapy (EET) in patients positive only on Seattle biopsy protocol for low-grade dysplasia (LGD), high-grade dysplasia (HGD), or esophageal adenocarcinoma (EAC) compared to proportion of patients referred for EET in patients positive only on WATS3D. All positive results for intestinal metaplasia/dysplasia or EAC with WATS3D sampling not detected on Seattle biopsy protocol at index endoscopy will require confirmation by repeat sampling using the Seattle biopsy protocol.
Interobserver agreement among pathologists for WATS3D specimens (Surveillance population only) | up to 6 months
  Interobserver agreement among pathologists with be assessed using Kappa statistics.
Predictors of dysplasia in patients with non-dysplastic BE (Surveillance population only) | up to 5 years
  Clinical and endoscopic variables collected as a part of the SWAT-BE study will be utilized to identify predictors associated with increased risk of progression to dysplasia or esophageal adenocarcinoma (EAC).
Counts of participants with a biomarker or panel of biomarkers associated with increased risk of progression | up to 5 years
  Specimens collected during the SWAT-BE study (WATS3D specimens) will be analyzed for biomarkers for improved risk stratification (i.e., identify patients at increased risk of progression to high-grade dysplasia or esophageal adenocarcinoma).
Diagnostic yield of dysplasia (Screening population only) | up to 1 year
  Proportion of positive results between the Seattle protocol and WATS3D technique. Positive results include low-grade dysplasia (LGD), high-grade dysplasia (HGD), and esophageal adenocarcinoma (EAC). All positive results for dysplasia or EAC with WATS3D sampling not detected on Seattle biopsy protocol at index endoscopy will require confirmation by repeat sampling using the Seattle biopsy protocol.

CONTACTS AND LOCATIONS:
Overall Officials: Sachin Wani, MD, Principal Investigator — University of Colorado, Denver
Locations (14):
- United States (14):
  - Arizona Centers of Digestive Health, Gilbert, Arizona
  - UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California
  - Kaiser Permanente, Oakland, California
  - University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - Connecticut Clinical Research Institute, Bristol, Connecticut
  - Suncoast Endoscopy of Sarasota, Sarasota, Florida
  - Northwestern University, Chicago, Illinois
  - Mayo Clinic, Rochester, Minnesota
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - Weill Cornell Medicine, New York, New York
  - University of Rochester, Rochester, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Geisinger Medical Center, Danville, Pennsylvania
  - Gastrointestinal Associates, PC, Knoxville, Tennessee

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in original publications after deidentification (text, tables, figures, appendixes).
Supporting Information: Study Protocol
Time Frame: 9 months to 36 months following article publication.
Access Criteria: Researchers who provide a methodologically sound proposal and investigators whose proposed use of the data has been approved by an independent review committee identified for this purpose.
  These data can only be used for individual participant data meta-analysis.